CLINICAL TRIAL: NCT06151899
Title: The Effect of Applying Kinesio Tape on Back Pain, Breastfeeding Success and Breastfeeding Self-Efficacy Levels in Mothers: Randomized Controlled Trial
Brief Title: Effect of Kinesio Tape on Back Pain, Breastfeeding Success and Breastfeeding Self-Efficacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Collaborators: Niğde Ömer Halisdemir University (Unknown); Selcuk University (Other)
Responsible Party: Principal Investigator, Merve Arı, M.Sc., KTO Karatay University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: ari1
Record Dates: First submitted 2023-10-26; First posted 2023-11-30 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Mothers Who Have Babies Between 0-6 Months and Are Actively Breastfeeding; Mothers Who Complain of Back Pain Due to Breastfeeding (Getting 6 Points or More on VAS in the Mothers' Own Evaluation)
Keywords: Pain; Breastfeeding; Breast milk; Nursing; Therapy
MeSH Terms: conditions — Pain; Breast Feeding

STUDY DESIGN:
Intervention Model Description: After the study is explained to mothers who meet the inclusion criteria and agree to participate in the study, their signatures on informed consent forms will be taken. Randomization will be random assignment to a control group or two intervention groups (1:1) with sequentially numbered, sealed, opaque envelopes containing randomly generated numbers after mothers have obtained informed consent. Randomization will be carried out via www.random.org using a table of random numbers.
Who Masked: Participant
Masking Description: Single (Participant)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio tape applying group (Experimental): To the mothers in the experimental group; Kinesio tape application will be performed by two experienced physiotherapists, one of whom is an expert and the other has a doctorate degree, with a kinesio tape certificate.
  Interventions: Other: Kinesio taping with angle and tension
- Control group (No Intervention): The control group will receive placebo kinesio taping.

INTERVENTIONS:
Other: Kinesio taping with angle and tension — Kinesio taping by applying angle and tension to back muscle
  Arms: Kinesio tape applying group

SUMMARY:
Back pain caused by posture changes and increased weight on the breasts during breastfeeding may negatively affect breastfeeding success and self-efficacy. Kinesio tape application, which is an effective and cost-effective method, can provide a more comfortable breastfeeding experience by controlling this pain.

DETAILED DESCRIPTION:
Despite the universality of these globally valid recommendations for the promotion of breastfeeding, the frequency and prevalence of breastfeeding rates vary from country to country and even between regions within certain countries. Planning and successful implementation of interventions to promote breast milk is possible by controlling both positive and negative factors that affect the success and duration of breastfeeding. In order to control the physical problems associated with breastfeeding, existing approaches in the literature for pain management such as fullness of the breasts due to increased lactation, poor positioning during breastfeeding, backaches. Kinesio taping is one of these methods, and since it does not have any pharmacological content, it is a practice that does not have side effects on breastfeeding and lactation.

ELIGIBILITY:
Inclusion Criteria:

* Mothers who have babies between 0-6 months and are actively breastfeeding
* Primiparous mothers
* Mothers who complain of back pain due to breastfeeding (Getting 6 points or more on VAS in the mothers' own evaluation)

Exclusion Criteria:

* Mothers with premature babies or babies with congenital anomalies
* Mothers taking painkillers
* Mothers diagnosed with posture disorders or skeletal system disorders
* Mothers whose breastfeeding is contraindicated
* Mothers whose breast milk has stopped
* Mothers who have other pain complaints in addition to back pain (such as nipple cracks, mastitis pain, etc.)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Active breastfeeding women
Enrollment: 60 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
The first outcome measure of the study is to examine the effect of Kinesio tape application on back pain in the mothers in the experimental group. | Average 2 weeks
  The VAS pain scale will be used for this.Visual Analog Scale (VAS): The scale is used to measure pain intensity. The scale consists of a 10 cm or 100 mm long horizontal or vertical ruler showing "no pain" at one end and "the most severe pain" possible at the other end. At the left end of the line is the expression "No pain" or "Pain is completely gone", while at the right end is the expression "Unbearable pain" or "There is no decrease in pain". A score of 6 and above indicates that the pain level has increased.
Mother Introduction Form | Average 2 weeks
  This form was prepared by the researchers in line with the literature. The form consists of 9 questions that question about breastfeeding process and her baby' demographics.

SECONDARY OUTCOMES:
The second outcome measure of the study is to determine the effect of the interventions on the breastfeeding success perception of the mothers in the experimental group. | Average 2 weeks
  1. LATCH Breastfeeding Diagnosis and Evaluation Scale: LATCH Breastfeeding Diagnosis Scale: L; Latch on the breast A; seeing/hearing the baby's swallowing movement (Audible swallowing) T; Type of the nipple C; comfort of the mother's breast and nipple (Comfort breast/nipple) H; It is the holding position of the baby (Hold/Help). A Turkish reliability study of the tool was conducted by Yenal and Okumuş, and it was found to be a suitable and reliable diagnostic tool for use. Each item is worth 0-2 points and the total score is a maximum of 10 points. A lower score indicates a need for support in breastfeeding.
The second outcome measure of the study is to determine the effect of the interventions on the breastfeeding self-efficacy of the mothers in the experimental group. | Average 2 weeks
  2. Breastfeeding Self-Efficacy Scale (EÖS): The minimum score that can be obtained from the scale is 14 and the maximum score is 70. A higher score indicates higher breastfeeding self-efficacy. The Turkish validity and reliability study of the scale was conducted by Tokat and Okumuş.

CONTACTS AND LOCATIONS:
Overall Officials: Hilal Kurt Sezer, Ph.D., Study Director — Nigde Omer Halisdemir University; Sibel Kucukoglu, Ph.D., Study Chair — Selcuk University; B. Sonmez Unuvar, Ph.D., Study Director — KTO Karatay University; Merve A. Ceran, Study Director — KTO Karatay University
Locations (1):
- KTO Karatay University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hay G, Baerug AB. The benefits of exclusive breastfeeding up to six months. Tidsskr Nor Laegeforen. 2019 May 3;139(9). doi: 10.4045/tidsskr.19.0105. Print 2019 May 28. No abstract available. English, Norwegian. PMID 31140258
- [Result] Admasu J, Egata G, Bassore DG, Feleke FW. Effect of maternal nutrition education on early initiation and exclusive breast-feeding practices in south Ethiopia: a cluster randomised control trial. J Nutr Sci. 2022 May 30;11:e37. doi: 10.1017/jns.2022.36. eCollection 2022. PMID 35720173
- [Result] Schafer EJ, Campo S, Colaizy TT, Mulder PJ, Breheny P, Ashida S. First-time mothers' breast-feeding maintenance: role of experiences and changes in maternal perceptions. Public Health Nutr. 2017 Dec;20(17):3099-3108. doi: 10.1017/S136898001700221X. Epub 2017 Sep 7. PMID 28879823
- [Result] Kucukoglu S, Sezer HK, Dennis CL. Validity and reliability of the Turkish version of the paternal breastfeeding self-efficacy scale - Short form for fathers. Midwifery. 2023 Jan;116:103513. doi: 10.1016/j.midw.2022.103513. Epub 2022 Oct 22. PMID 36323075
- [Result] Lambrinou CP, Karaglani E, Manios Y. Breastfeeding and postpartum weight loss. Curr Opin Clin Nutr Metab Care. 2019 Nov;22(6):413-417. doi: 10.1097/MCO.0000000000000597. PMID 31577639
- [Result] Lockyer F, McCann S, Moore SE. Breast Milk Micronutrients and Infant Neurodevelopmental Outcomes: A Systematic Review. Nutrients. 2021 Oct 28;13(11):3848. doi: 10.3390/nu13113848. PMID 34836103
- [Result] Milinco M, Travan L, Cattaneo A, Knowles A, Sola MV, Causin E, Cortivo C, Degrassi M, Di Tommaso F, Verardi G, Dipietro L, Piazza M, Scolz S, Rossetto M, Ronfani L; Trieste BN (Biological Nurturing) Investigators. Effectiveness of biological nurturing on early breastfeeding problems: a randomized controlled trial. Int Breastfeed J. 2020 Apr 5;15(1):21. doi: 10.1186/s13006-020-00261-4. PMID 32248838
- [Result] Anderson L, Kynoch K, Kildea S, Lee N. Effectiveness of breast massage for the treatment of women with breastfeeding problems: a systematic review. JBI Database System Rev Implement Rep. 2019 Aug;17(8):1668-1694. doi: 10.11124/JBISRIR-2017-003932. PMID 31135656
- See also: WHO — https://www.who.int/publications/i/item/9789241565707